CLINICAL TRIAL: NCT06334484
Title: Effect of Advanced Hybrid Closed Loop System on Adjunctive Continuous Glucose Monitoring Metrics, Two-years Observational Study
Brief Title: Effect of Advanced Hybrid Closed Loop System on Adjunctive Continuous Glucose Monitoring Metrics
Acronym: TiTR_GR1DM
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6413
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Advanced hybrid closed loop systems — Collect data from advanced hybrid closed loop users

SUMMARY:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease characterized by pancreatic beta cells destruction, resulting in insulin secretion deficit (1). Insulin therapy is essential in the therapeutical management of subjects with T1DM (1). The Diabetes Complications and Control Trial (DCCT) has showed that intensive insulin treatment was associated with a reduction in the onset of complications related to diabetes. In recent years, treatment of T1DM evolved rapidly because of the significant improvements in the use of technology (2). With the spread of continuous glucose monitoring (CGM) systems, standardized metrics, summarizing time spent within optimal glucose range (time in range - TIR), time below target glucose range (TBR) and time above target glucose range (TAR), have become commonly used metrics in clinical practice (3,4). Furthermore, glucose management indicator (GMI) estimates glycated haemoglobin from the average glucose level of CGM readings for 14 days and coefficient of variation (CV) evaluates the amplitude of glucose excursions.

Advanced hybrid closed loop (AHCL) systems combine insulin pump infusion and real time CGM (rtCGM) data through an algorithm: they suspend insulin infusion if hypoglycaemia is expected and can administer automatic corrective boluses in case of hyperglycaemia (6). Different algorithms, as Model Predictive Control (MPC) or Proportional-Integral-Derivative (PID), are used by different systems available on the market and are currently used in clinical practice. Overall, AHCL are associated with improvement of glycated hemoglobin (HbA1c) and TIR opening to the possibility to gain even tighter glycemic control.

The primary objective is therefore to evaluate the glycemic improvement expressed through adjunctive CGM metrics in subjects with T1DM 24 months after starting AHCL therapy

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed before any activity related to the study
2. Age ≥18 years, both sexes
3. Start of AHCL for at least 6 months before enrollment (from 01/01/2021 to 31/12/2023).

Exclusion Criteria:

1. Diagnosis of type 2 diabetes mellitus or other forms of diabetes, such as metasteroid diabetes, secondary to pancreatectomy, related to pancreatitis or secondary to endocrinological disorders, gestational diabetes, maturity-onset diabetes of the young (MODY).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with T1DM who started AHCL for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2025-09-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
change in time spent in tighter glucose range after 24 months of hybrid closed loop system | 24 months
  time spent in tighter glucose range (TiTR - 70-140 mg/dl or 3.9-7.8 mmol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy